CLINICAL TRIAL: NCT00908089
Title: Use of TNF-blocking Therapy in Combination With DMARDs in Patients With Early Rheumatoid Arthritis
Brief Title: TNF-blocking Therapy in Combination With Disease-modifying Antirheumatic Drugs in Early Rheumatoid Arthritis
Acronym: NEO-RACo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Seinajoki Central Hospital (Other); Oulu University Hospital (Other); Jyväskylä Central Hospital (Other); Kuopio University Hospital (Other); Satakunta Central Hospital (Other); University of Turku (Other); Rheumatism Foundation Hospital (Other); Orton Invalid Foundation (Other); South Carelia Central Hospital (Other); Lappi Central Hospital (Unknown); Kanta-Häme Central Hospital (Other Government)
Responsible Party: Principal Investigator, Marjatta Leirisalo-Repo, MD, PhD, Prof, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEO-RACo
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; methotrexate; sulfasalazine; hydroxychloroquine; infliximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Naltrexone; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trexan+Salazopyrin+Oxiklorin+prednisolone + infliximab (Active Comparator): Combination therapy with 3 DMARDs (starting with methotrexate 10-25 mg/week, sulphasalazine 1-2 g/day and hydroxychloroquine 35 mg/kg/week)+ Prednisolon 7.5 mg/day + infliximab 3 mg/kg at weeks 4, 6, 10, 18, 26
  Interventions: Drug: Trexan+Salazopyrin+Oxiklorin+prednisolone + infliximab
- Trexan+Salazopyrin+Oxiklorin+prednisolone + placebo (Placebo Comparator): Combination therapy with 3 DMARDs (starting with methotrexate 10-25 mg/week, sulphasalazine 1-2 g/day and hydroxychloroquine 25 mg/kg/week)+ Prednisolon 7.5 mg/day + placebo at weeks 4, 6, 10, 18, 26
  Interventions: Drug: Trexan+Salazopyrin+Oxiklorin+prednisolone + placebo

INTERVENTIONS:
Drug: Trexan+Salazopyrin+Oxiklorin+prednisolone + infliximab — methotrexate 10-25 mg/week, sulfasalazine 1-2 g/day, hydroxychloroquine 35 mg/kg/week, prednisolone 7.5 mg/day, and infliximab 3 mg/kg during first 6 months
  Other Names: Trexan, Salazopyrin, Oxiklorin, Prednison, Remicade
  Arms: Trexan+Salazopyrin+Oxiklorin+prednisolone + infliximab
Drug: Trexan+Salazopyrin+Oxiklorin+prednisolone + placebo — methotrexate 10-25 mg/week, sulfasalazine 1-2 g/day, hydroxychloroquine 35 mg/kg/week, prednisolone 7.5 mg/day, and placebo infusion during first 6 months
  Other Names: Trexan, Salazopyrin, Oxiklorin, Prednison, 0.9% NaCl
  Arms: Trexan+Salazopyrin+Oxiklorin+prednisolone + placebo

SUMMARY:
The FIN-RACo trial is an investigator initiated multicenter (n=15 centers in Finland) prospective study on the treatment of patients with early rheumatoid arthritis (RA) with combination therapy with disease modifying antirheumatic drugs starting with methotrexate, sulphasalazine, hydroxychloroquine and prednisolone (COMBI). During the first 6 months, the patients are randomized to treatment with infliximab/placebo added on the combination treatment. The study is prospective for 5 years, with extension to 10 years. The target is to induce remission in both treatment arms. To reach this target, the investigators use frequent changes of doses and anti-rheumatic drugs and use of intra-articular glucocorticoid injections. The primary endpoints are the proportions of patients with remission at 2 and 5 years in both treatment arms.

DETAILED DESCRIPTION:
We want to study, whether early treatment with infliximab for 6 months started parallel with the combination therapy of methotrexate, sulphasalazine, hydroxychloroquine and prednisolone (COMBI) can induce quick remission in patients with early RA, if the remission can be sustained after 6 months on patients continuing the COMBI treatment and can diminish the risk of progression of erosive changes in patients with early RA, and if we can reduce costs of the 2 treatment arms with respect to costs due to the disease.

100 patients with early RA will be included in the study. The patients are randomised into COMBI + placebo or into COMBI +infliximab.

All patients are treated openly with COMBI, starting with a combination of methotrexate, sulfasalazine, hydroxychloroquine and prednisolone. In addition, the patients are randomized into a) infliximab or b) similar placebo. The COMBI treatment will be continued for 2 years, but the infliximab/placebo will be given only during the first 6 months. After 2 years, if the patient is in remission, the prednisolone will be gradually tapered off. If the patient is still in remission, the conventional DMARDs can be sequentially tapered down. If the remission is lost, the last DMARD is reinstituted. If the patient is not in remission of COMBI, after 26 weeks, treatments are free, including the institution of a biological drug.

The patients will be evaluated clinically at week 0, 4, 6, 10, 14, 18, 22 and 26 (at the day of infusion, prior to the infusion) and at months 8, 10, 12, 15, 18, 21, and 24 and at annually thereafter till 10 years.

If a patient has adverse events due to individual drugs in the COMBI, the treatment can be substituted by another DMARD.The disease activity will be measured according to the ACR core set of disease activity.

Radiology of hands (PA projection) and feet (PA projection) at baseline and at 1, 2, 3, 4, 5, 7 and 10 years. We also will record adverse events, sick leaves, loss of income, costs, and work disability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA fulfilling the ACR classification criteria for RA
* Patients within age group of 18-60 years
* Patients not permanently work disabled or retired
* Duration of symptoms < 12 months, and who have not received DMARD previously
* Patients with active disease (see below)
* Criteria for active disease at entry:

  * > 6 swollen joints (66 joint count)
  * > 6 tender joints (68 joint count)
  * duration of early morning stiffness > 45 min and/or ESR > 30 mm/h and/or CRP > 20 mg/l

Exclusion Criteria:

* Previous treatment with DMARDs
* Previous treatment with oral glucocorticoids during the previous 6 months
* Less than 30 days from previous intra-articular injection with corticosteroids
* Allergy to sulphonamides
* Allergy to acetylsalicylic acid
* Allergy to methotrexate
* Allergy to antimalarials
* Previous treatment with biologicals
* Serum creatinine value > upper limit of normal (registered in 2 different blood samples)
* Serum transaminase levels > 2x upper limit of normal (registered in 2 different samples)
* Known/previous malignancy excluding basalioma or in situ cervical cancer >5 years previously
* Cardiac failure (NYHA III-IV)
* Previous history of tuberculosis and/or exposition to tuberculosis and/or typical changes of previous/active tuberculosis in chest radiology
* Active infection
* Pregnancy
* Leukopenia (WBC < 4 x 109/l)
* Thrombocytopenia (platelets < 100 x 109/l)
* Active peptic ulcer
* Type I or type II diabetes under poor control
* Heavy use of alcohol
* Fertile women not practising contraception or who are planning pregnancy
* Male patients wishing to have children during the therapy
* Other autoimmune rheumatic disease
* Other chronic disease which judged by the physician could influence the patient's compliance or intervene the study course
* Patient is not cooperative

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2003-03; Primary Completion 2007-05 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Remission by ACR criteria | 2 years

SECONDARY OUTCOMES:
Radiology (erosions) | 2 years
Sustained remission | 2 years
  Number of patients with sustained ACR remission from month 3 till the end of the study
Costs | 2
  Cumulative direct and indirect costs at 2 years

OTHER OUTCOMES:
HAQ | 1, 2, 3, 4 and 5 years
  Health assessment questionnaire(HAQ)
Work disability | 2, 3, 4 and 5 years
  Permanent work disability
Good response | 5 years
  Number of patients with sustained good response (>=ACR50%) from month 3 till the end of study
Number of arthroplasties | 5 years
  Cumulative number of arthroplasties at 5 years
Direct and indirect costs | 5 years
  Cumulative direct an indirect costs at 5 years
Adverse events | 10 years
  Monitoring of safety and adverse events
ACR Remission | 10 years
DAS28 remission | 2, 3, 4, 5, 7 and10 years
HAQ | 10 years
  Health assessment questionnaire (HAQ)
Work disability | 10 years
  Cumulative permanent work disability up till 10 years
Number of arthroplasties | 10 years
  Cumualite number of arthroplasties by 10 years
Direct and indirect costs | 10 years
  Cumulative direct and indirect costs by 10 years
Radiology (erosions) | 10 years
  radiologic changes in hands and feet

CONTACTS AND LOCATIONS:
Overall Officials: Marjatta Leirisalo-Repo, MD, Prof, Study Director — University of Helsinki; Timo Möttönen, MD, Prof, Study Chair — University of Turku; Markku Korpela, MD, PhD, Study Chair — Tampere University; Riitta Luosujärvi, MD, PhD, Study Chair — Helsinki University Central Hospital; Oili Kaipiainen-Seppänen, MD, PhD, Study Chair — Kuopio University Hospital; Markku Kauppi, MD, PhD, Study Chair — Päijänne Tavastia Central Hospital
Locations (13):
- Finland (13):
  - Hämeenlinna Central Hospital, Hämeenlinna
  - Rheumatism Foundation Hospital, Heinola
  - Helsinki University Central Hospital, Helsinki
  - Orton Invalid Foundation Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Lappeenranta Central Hospital, Lappeenranta
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Rauma
  - Rovaniemi Central Hospital, Rovaniemi
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku

REFERENCES:
- [Result] Leirisalo-Repo M, Kautiainen H, Laasonen L, Korpela M, Kauppi MJ, Kaipiainen-Seppanen O, Luosujarvi R, Luukkainen R, Karjalainen A, Blafield H, Uutela T, Ilva K, Julkunen HA, Paimela L, Puolakka K, Moilanen E, Hannonen PJ, Mottonen T; NEO-RACo Study Group. Infliximab for 6 months added on combination therapy in early rheumatoid arthritis: 2-year results from an investigator-initiated, randomised, double-blind, placebo-controlled study (the NEO-RACo Study). Ann Rheum Dis. 2013 Jun;72(6):851-7. doi: 10.1136/annrheumdis-2012-201365. Epub 2012 Jun 30. PMID 22753402
- [Result] Rantalaiho V, Kautiainen H, Jarvenpaa S, Korpela M, Malmi T, Hannonen P, Kaipiainen-Seppanen O, Yli-Kerttula T, Mottonen T, Mustila A, Karjalainen A, Paimela L, Uutela T, Leirisalo-Repo M; NEO-RACo Study Group. Failure in longterm treatment is rare in actively treated patients with rheumatoid arthritis, but may be predicted by high health assessment score at baseline and by residual disease activity at 3 and 6 months: the 5-year followup results of the randomized clinical NEO-RACo trial. J Rheumatol. 2014 Dec;41(12):2379-85. doi: 10.3899/jrheum.140267. Epub 2014 Oct 1. PMID 25274892
- [Result] Rantalaiho V, Kautiainen H, Korpela M, Hannonen P, Kaipiainen-Seppanen O, Mottonen T, Kauppi M, Karjalainen A, Laiho K, Laasonen L, Hakola M, Peltomaa R, Leirisalo-Repo M; NEO-RACo Study Group. Targeted treatment with a combination of traditional DMARDs produces excellent clinical and radiographic long-term outcomes in early rheumatoid arthritis regardless of initial infliximab. The 5-year follow-up results of a randomised clinical trial, the NEO-RACo trial. Ann Rheum Dis. 2014 Nov;73(11):1954-61. doi: 10.1136/annrheumdis-2013-203497. Epub 2013 Aug 1. PMID 23908187
- [Derived] Sandstrom T, Kaipiainen-Seppanen O, Mali M, Kauppi M, Kautiainen H, Hannonen P, Yli-Kerttula T, Leirisalo-Repo M, Rantalaiho V. Limited reduction of bone mineral density in patients with early rheumatoid arthritis receiving aggressive treatment: 10 year results of the NEO-RACo study. Scand J Rheumatol. 2025 Nov;54(6):412-420. doi: 10.1080/03009742.2025.2515696. Epub 2025 Jun 23. PMID 40548492
- [Derived] Vuolteenaho K, Tuure L, Nieminen R, Laasonen L, Leirisalo-Repo M, Moilanen E; NEO-RACo Study Group. Pretreatment resistin levels are associated with erosive disease in early rheumatoid arthritis treated with disease-modifying anti-rheumatic drugs and infliximab. Scand J Rheumatol. 2022 May;51(3):180-185. doi: 10.1080/03009742.2021.1929456. Epub 2021 Jul 15. PMID 34263700
- [Derived] Sandstrom T, Rantalaiho V, Yli-Kerttula T, Kautiainen H, Malmi T, Karjalainen A, Uusitalo T, Julkunen H, Kaipiainen-Seppanen O, Paimela L, Puolakka K, Uutela T, Mottonen T, Hannonen P, Leirisalo-Repo M, Laasonen L, Kauppi M; NEO-RACo Study Group. Cervical Spine Involvement among Patients with Rheumatoid Arthritis Treated Actively with Treat-to-target Strategy: 10-year Results of the NEO-RACo Study. J Rheumatol. 2020 Aug 1;47(8):1160-1164. doi: 10.3899/jrheum.190139. Epub 2019 Nov 15. PMID 31732558
- [Derived] Rantalaiho V, Sandstrom T, Koski J, Hannonen P, Mottonen T, Kaipiainen-Seppanen O, Yli-Kerttula T, Kauppi MJ, Uutela T, Malmi T, Julkunen H, Laasonen L, Kautiainen H, Leirisalo-Repo M; NEO-RACo Study Group. Early Targeted Combination Treatment With Conventional Synthetic Disease-Modifying Antirheumatic Drugs and Long-Term Outcomes in Rheumatoid Arthritis: Ten-Year Follow-Up Results of a Randomized Clinical Trial. Arthritis Care Res (Hoboken). 2019 Nov;71(11):1450-1458. doi: 10.1002/acr.23782. PMID 30295425